CLINICAL TRIAL: NCT01828879
Title: The Efficacy and Safety of Tacrolimus Ointment in Adult Patients With Moderate to Severe Atopic Dermatitis
Brief Title: An Efficacy and Safety Study of Tacrolimus Ointment in Adult Participants With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Ltd.,Thailand (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017833; R098924ADM4006
Record Dates: First submitted 2013-03-21; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Dermatitis, Atopic
Keywords: Dermatitis, Atopic; Tacrolimus
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus ointment (Experimental): Tacrolimus ointment, 0.1 percent will be applied twice daily, in adult population for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first.
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus ointment, 0.1 percent will be applied twice daily, in adult population for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of tacrolimus ointment in treating the signs and symptoms of moderate (medium level of seriousness) to severe (very serious, life threatening) atopic dermatitis (an intensely pruritic [itching], chronic [lasting a long time], inflammatory [pain and swelling], immunologically based skin disease with a genetic predisposition [latent susceptibility to disease at the genetic level]) in adult participants.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), prospective (study following participants forward in time), randomized (like the flip of a coin), multi-center study in adult participants with moderate to severe atopic dermatitis. Participants will be treated with 0.1 percent concentration of tacrolimus ointment which will be applied twice daily for 4 weeks or until 1 week after the affected areas defined for treatment at baseline are completely cleared, whichever is first. The study will consist of 6 visits: pre-study (optional), Baseline or Day 1, Weeks 1, 2, 3 and 4 (end-of-treatment). The ointment should be applied at least 2 hours before or at least 30 minutes after bathing, showering, shaving, use of sauna, or heavy exercise (i.e. causes sweating). On study visit days, the ointment should be applied at least 2 hours before the visit. Efficacy evaluation will be done at all subsequent study visits in participants receiving study drug for at least 3 consecutive days (minimum of 5 applications) while the participants who will receive at least 1 application of the study drug, will be evaluated for safety. Primary efficacy evaluation will be based on the Physician's Global Evaluation of Clinical Response (PhGECR). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of atopic dermatitis using Hanifin and Rajka Criteria (major criteria: pruritus, lichenification [crusting over], chronic relapsing [the return of a medical problem] course, family history of atopy and minor criteria: xerosis [dry skin], ichthyosis [skin disorders characterized by dryness, roughness, and scaliness], immediate Type I reactions [reactions which occur within minutes of exposure to challenging antigen: substances that are recognized by the immune system and induce an immune reaction] to skin test antigens) involving at least 10 percent of the body surface area
* Participants not having other skin disorders and severe heart, liver, kidney and lung diseases
* Participants who have given informed consent
* Female participants with child-bearing potential must have a negative pregnancy test
* Participant meets the following washout requirements (washout period ranging from 1-42 days) before study: 1 day (for non-medicated topical [applied to skin; surface] agents); 7 days (for terfenadine, other non-sedating systemic antihistamines [drug used to treat allergic reaction], topical corticosteroids (steroid hormone), H1 and H2 antihistamines, antimicrobial [drug that kills bacteria and other germs], other medicated topical agents); 14 days (for intranasal [delivery of medications through the nasal mucosa] and/or inhaled corticosteroids); 28 days (for light treatments [ultra violet rays A, ultra violet rays B], non-steroidal immunosuppressants [drug which suppresses the body's immune response, used in transplantation and diseases caused by disordered immunity], other investigational drugs and systemic corticosteroids); and 42 days (for astemizole)

Exclusion Criteria:

* Participant with a skin disorder other than atopic dermatitis in the areas to be treated
* Participant who have pigmentation or extensive scarring or pigmented lesions (abnormal area of tissue, such as a wound, sore, rash, or boil) in the areas to be treated which would interfere with rating of efficacy parameters
* Participant who have clinically infected atopic dermatitis at baseline
* Participant with a systemic disease, including cancer (abnormal tissue that grows and spreads in the body until it kills) or a history of cancer or Human Immunodeficiency Virus (HIV: a life-threatening infection which you can get from an infected person's blood or from having sex with an infected person), which would contraindicate (medical reasons that prevent a person from using a certain drug or treatment) the use of immunosuppressants
* Participant with a known hypersensitivity (altered reactivity to an antigen) to macrolides (drugs exhibiting antibiotic properties) or any excipient of the ointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2007-11; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Physician's Global Evaluation of Clinical Response (PhGECR) | Week 4
  PhGECR scale evaluates the change in the lesions of atopic dermatitis, which is defined as the lesions identified by Investigator for treatment at Baseline only, using scores ranging from, less than 0 to 100: wherein, less than 0=worse, 0-29=no appreciable improvement, 30-49=slight improvement, 50-74=moderate improvement, 75-89=marked improvement, 90-99=excellent improvement and 100=cleared.

SECONDARY OUTCOMES:
Eczema Area and Severity Index (EASI) | Week 1, 2, 3 and 4
  A composite index of area involved and severity of the signs of atopic dermatitis in the 4 regions (head and neck, upper limbs, trunk, lower limbs) will be calculated using the physician's assessment of individual signs using a scale ranging from 0 to 3: 0=absent, 1=mild, 2=moderate, 3=severe; and the affected area assessment (the percentage of body surface area affected by atopic dermatitis) of the lesions defined in the baseline treatment area will be estimated by the physician on the basis of area score ranging from 0 to 6: 0=0 percent and 6=90 to 100 percent.
Participant's Assessment of Treatment Effects | Week 1, 2, 3 and 4
  Participants will make 2 assessments at each study visit (before and after treatment) based on all affected areas (ratio of 100 percent). The assessment rates include: much better, better, slightly better, same, slightly worse, worse. Much better and better is considered good.
Participant's Assessment of Itch | Week 1, 2, 3 and 4
  Participant's itch will be assessed using a Visual Analog Scale ranging from 0 to 100: 0-19=no or slight itch; 20-39=mild itch; 40-59=moderate itch; 60-79=severe itch; 80-100=worst itch.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd.,Thailand Clinical Trial, Study Director — Janssen-Cilag Ltd.,Thailand
Locations (2):
- Vietnam (2):
  - Hanoi
  - Hochiminh

REFERENCES:
- See also: The efficacy and safety of tacrolimus ointment in Adult patients with moderate to severe atopic dermatitis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2487&filename=CR017833_CSR.pdf